CLINICAL TRIAL: NCT00231465
Title: Phase II Study of Taxotere® (Docetaxel) + ZD1839 (IRESSA®) in Previously Untreated Elderly Patients (≥70 Years Old) With Stage III-b (With Malignant Pleural Effusion [MPE+]) or Stage IV Non-Small Cell Lung Cancer (NSCLC)
Brief Title: Phase II Study of Docetaxel + ZD1839 in Elderly Patients With Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-12905; 1839US/0205 (Other: AstraZeneca)
Record Dates: First submitted 2005-10-03; First posted 2005-10-04 (Estimated); Results first posted 2012-11-30 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2012-08

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: elderly; malignant pleural effusion
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Pleural Effusion, Malignant | interventions — Docetaxel; Gefitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Taxotere® (Docetaxel) + ZD1839 (IRESSA®) (Experimental): Patients will receive Taxotere at 75 mg/m2 given IV over 60 minutes on day 1 of a three week cycle.
  ZD1839 will be administered orally at 250mg daily starting on day one, concurrently with the Taxotere.
  Interventions: Drug: docetaxel (Taxotere®); Drug: ZD1839

INTERVENTIONS:
Drug: docetaxel (Taxotere®) — Taxotere® will be administered to patients a maximum of 2 cycles, after a maximal response is achieved, and then discontinued.
  Other Names: Taxotere®
Drug: ZD1839 — ZD1839 will be continued until progression, or until trial closure, whichever comes first.
  Other Names: IRESSA®; gefitinib

SUMMARY:
This is a Phase II, open-label trial of Taxotere® + ZD1839 in elderly patients with Stage III-b or IV NSCLC who have received no prior chemotherapy for metastatic disease. Patients with prior adjuvant chemotherapy were allowed to enroll on this trial.

DETAILED DESCRIPTION:
This trial is designed to test the efficacy and tolerability of a standard chemotherapy agent, Docetaxel, in combination with an oral agent, Iressa, in elderly patients with advanced stage lung cancer. Current practices utilize two chemotherapeutic medications that may result in increased toxicities and poor outcomes in the elderly population. Treatment consists of an infusion of docetaxel every 21 days for four doses while taking Iressa every day. A computed tomography (CT) scan will measure disease response after two cycles. Response determines continuation of treatment. Lab work will be collected before every treatment. Side effect information will also be collected at every visit. Once the infusion phase of the study is completed, a maintenance phase of taking just the Iressa begins and disease assessment occurs every two months. This period will last until disease progression is demonstrated.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be greater than or equal to 70 years of age.
* Patients must have histologically confirmed non-small cell lung cancer (NSCLC) that is Stage IIIb (with pleural effusions) or Stage IV.
* Patients must be previously untreated for metastatic disease but may have received previous adjuvant chemotherapy more than six months prior to registration. Patients may also have received radiation therapy for advanced disease; however there should be measurable disease outside the radiation ports.
* Disease must be at least unidimensionally measurable. Lesions, which are located within a previously irradiated field, are not considered measurable unless there is a documented growth in its size.
* Patients must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Laboratory values must be as follows: White blood cell count greater than or equal to 3,000/mm^3; Absolute neutrophil count greater than or equal to 1,500/mm^3; Platelets greater than or equal to 100,000/mm^3; Total bilirubin less than or equal to 1.0 x institutional upper normal limit; Serum creatinine less than or equal to 2 x institutional upper normal limit; aspartic transaminase (AST) or ALANINE TRANSAMINASE (ALT) less than or equal to 1.5 x institutional upper normal limit; Alkaline Phosphatase less than or equal to 1.5 x institutional upper normal limit; Serum calcium less than or equal to 1.5 x institutional upper normal limit (corrected for serum albumin).
* Patients with combined alkaline phosphatase, AST and/or ALT elevations will not be allowed to enroll on protocol.
* Patients must have recovered from all acute toxicities from previous therapy, excluding alopecia.
* In keeping with the policies of the institution, patients must sign an informed consent form indicating that they are aware of the investigational nature of this study
* Patients with stable brain metastases after completion of radiation will be allowed to enroll in this trial.
* Patients treated with adjuvant therapy more than six months ago will be allowed to enroll in this trial.
* Cognitively impaired patients will be allowed to enroll on the trial if the legal guardian signs the consent form after a full informed consent process is completed. Whenever feasible the cognitively impaired person will also give assent to participation in the trial.

Exclusion Criteria:

* Patients previously treated with chemotherapy or ZD1839.
* Patients with known or clinical evidence of active central nervous system (CNS) metastasis. Patients with stable, previously treated brain metastases will be allowed.
* Male Patients with female sexual partners in the reproductive age group who refuse to use effective methods of contraception will be excluded from the trial.
* Patients with concurrent serious infections (i.e., receiving an intravenous antibiotic) are not eligible.
* Patients with an unstable or serious concurrent medical condition are excluded. Examples include, but are not limited to, uncontrolled ventricular arrhythmia, recent (within 3 months) myocardial infarction, uncontrolled major seizure disorder, grade 3 neuropathies, spinal cord compression, superior vena cava syndrome, or any psychiatric disorder that prohibits obtaining informed consent.
* Patients receiving other non-approved or investigational therapy concurrently or within 30 days of Day 1 of trial treatment.
* Patients with a history of other cancers except basal cell skin cancers, carcinoma of the cervix in situ, or curatively-treated cancers with > 2 years non-recurrence prior to entry in the trial. Patients with a history of other cancers must have histological confirmation that current disease is compatible with diagnosis of NSCLC.
* Peripheral neuropathy >2. (Peripheral neuropathy must be < grade 1)
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to Docetaxel, ZD 1839, Polysorbate 80, or other agents used in the study.
* Patients with combined alkaline phosphatase, AST and/or ALT elevations will be excluded from this protocol.
* Patients previously treated with radiation therapy.

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 44 (Actual)
Dates: Start 2003-07; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alberto Chiappori, MD, Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center & Research Institute, Tampa, Florida, United States

REFERENCES:
- [Derived] Simon GR, Extermann M, Chiappori A, Williams CC, Begum M, Kapoor R, Haura EB, Ismail-Khan R, Schell MJ, Antonia SJ, Bepler G. Phase 2 trial of docetaxel and gefitinib in the first-line treatment of patients with advanced nonsmall-cell lung cancer (NSCLC) who are 70 years of age or older. Cancer. 2008 May 1;112(9):2021-9. doi: 10.1002/cncr.23360. PMID 18300255

RESULTS

PARTICIPANT FLOW:
Groups:
- Taxotere® (Docetaxel) + ZD1839 (IRESSA®): Eligible patients were treated with docetaxel 75 mg/m2 every three weeks and gefitinib 250 mg orally daily. Docetaxel and ZD1839 (gefitinib) were given for two cycles beyond maximal response. Gefitinib was continued until disease progression. Co-morbidities and activities of daily living were assessed (IADL).
Period: Overall Study
Arm/Group | Taxotere® (Docetaxel) + ZD1839 (IRESSA®)
Started | 44
Completed | 42
Not Completed | 2
Not completed — Completed only one cycle | 1
Not completed — Did not have follow up CT scans | 1

BASELINE CHARACTERISTICS:
Groups:
- Taxotere® (Docetaxel) + ZD1839 (IRESSA®): Patients will receive Taxotere at 75 mg/m2 given IV over 60 minutes on day 1 of a three week cycle.
  ZD1839 will be administered orally at 250mg daily starting on day one, concurrently with the Taxotere.
  ZD1839 : ZD1839 will be continued until progression, or until trial closure, whichever comes first.
  docetaxel (Taxotere®) : Taxotere® will be administered to patients a maximum of 2 cycles, after a maximal response is achieved, and then discontinued.
Arm/Group | Taxotere® (Docetaxel) + ZD1839 (IRESSA®)
Number analyzed (Participants) | 44
Age, Customized [Median (Full Range); unit: years] | 75 [70 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 26
Region of Enrollment [Number; unit: participants]
  United States | 44

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR)
Description: ORR: Complete Response (CR) + Partial Response (PR). Response rate for Elderly (> 70 years) previously untreated patients with Stage IIIb (With Malignant Pleural Effusion (MPE)) or IV non-small cell lung cancer (NSCLC) receiving Taxotere + ZD1839. Best clinical response to treatment with combination was determined using Response Evaluation Criteria in Solid Tumors (RECIST V1.0): * Complete Response (CR)- Disappearance of all target lesions; * Partial Response (PR)- At least a 30% decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum LD; * Progressive Disease (PD)- At least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions; * Stable Disease (SD)- Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum LD since the treatment started.
Time Frame: Duration of time on study, an average of 19 months
Population: Response was evaluable in 42 of the 44 patients.
Measure: Mean (95% Confidence Interval); unit: percentage of participants
Arm/Group | Taxotere® (Docetaxel) + ZD1839 (IRESSA®)
Number analyzed (Participants) | 42
percentage of participants | 40 [26 to 57]

2. Secondary Outcome: Progression Free Survival (PFS) Rate
Description: PFS was calculated from the date of enrollment to the date of progression. All 44 treated were assessed for PFS, with a minimum follow-up of 19 months. Progression (PD): At least a 20% increase in the sum of LD of target lesions taking as references the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions.
Time Frame: Duration of time on study, an average of 19 months
Population: All participants who initiated therapy between March 2003 and May 2005
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Taxotere® (Docetaxel) + ZD1839 (IRESSA®)
Number analyzed (Participants) | 44
Months | 6.9 [3.95 to 7.8]

3. Secondary Outcome: Overall Survival (OS) Rate
Description: OS was calculated from the date of enrollment to the date of death. All 44 treated were assessed for OS, with a minimum follow-up of 19 months.
Time Frame: Duration of time on study, an average of 19 months
Population: All participants who initiated therapy between March 2003 and May 2005
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Taxotere® (Docetaxel) + ZD1839 (IRESSA®)
Number analyzed (Participants) | 44
Months | 9.59 [4.6 to 16.3]

ADVERSE EVENTS:
Time Frame: 7 years, 2 months
Arm/Group | Taxotere® (Docetaxel) + ZD1839 (IRESSA®)
Serious Adverse Events (participants affected / at risk) | 14/44
Other Adverse Events (participants affected / at risk) | 38/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Taxotere® (Docetaxel) + ZD1839 (IRESSA®) (N=44)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Neutropenia (Infections and infestations) | 1 (1)
Lymphopenia (Blood and lymphatic system disorders) | 8 (8)
Febrile neutropenia (Infections and infestations) | 4 (4)
Hyperglycemia (Metabolism and nutrition disorders) | 5 (5)
Fatigue (General disorders) | 4 (4)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Elevated SGPT (Metabolism and nutrition disorders) | 2 (2)
Pulmonary Infiltrates (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 3 (3)
Dysphagia/Esophagitis (Gastrointestinal disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1)
Pneumonia (neutropenic) (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Exacerbation of COPD (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Elevated creatinine (Metabolism and nutrition disorders) | 1 (1)
Interstitial cystitis (Renal and urinary disorders) | 1 (1)
Syncope (General disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1)
Stroke (Vascular disorders) | 1 (1)
Herpes zoster (Infections and infestations) | 1 (1)
Dehydration (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Taxotere® (Docetaxel) + ZD1839 (IRESSA®) (N=44)
Neutropenia (Infections and infestations) | 4 (4)
Thrombocytopenia (Blood and lymphatic system disorders) | 4 (4)
Lymphopenia (Blood and lymphatic system disorders) | 32 (43)
Fatigue (General disorders) | 35 (60)
Alopecia (Skin and subcutaneous tissue disorders) | 24 (35)
Rash (Skin and subcutaneous tissue disorders) | 11 (11)
Hyperglycemia (Metabolism and nutrition disorders) | 6 (20)
Cough (Respiratory, thoracic and mediastinal disorders) | 15 (18)
Nail changes (Skin and subcutaneous tissue disorders) | 7 (7)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 15 (23)
Neuropathy - Sensory (Nervous system disorders) | 4 (4)
Bone pain (General disorders) | 3 (3)
Edema (Blood and lymphatic system disorders) | 4 (5)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 3 (3)
Nausea (Gastrointestinal disorders) | 3 (3)
Alkaline phosphatase (Blood and lymphatic system disorders) | 9 (22)
Anorexia (Metabolism and nutrition disorders) | 13 (15)
Fever (General disorders) | 2 (2)
Allergic rhinitis (Skin and subcutaneous tissue disorders) | 2 (3)
Bone Pain (General disorders) | 5 (5)
Constipation (Gastrointestinal disorders) | 5 (7)
Creatinine (Renal and urinary disorders) | 8 (29)
Diarrhea w/o colostomy (Gastrointestinal disorders) | 10 (17)
Dizziness (General disorders) | 3 (3)
Dry skin (Skin and subcutaneous tissue disorders) | 21 (35)
Dyspepsia (Gastrointestinal disorders) | 2 (3)
Dysphagia (Gastrointestinal disorders) | 3 (3)
Hemoglobin (Blood and lymphatic system disorders) | 25 (89)
Hypercalcemia (Metabolism and nutrition disorders) | 2 (2)
Stomatitis (Gastrointestinal disorders) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes